CLINICAL TRIAL: NCT03851536
Title: Transvaginal Versus Transabdominal Ultrasound Guided Embryo Transfer. Randomized Controlled Trial.
Brief Title: Ultrasound Guidance for Embryo Transfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Principal Investigator, Haitham Aboali Hamza, Lecturer of Obstetrics and Gynecology, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU179
Record Dates: First submitted 2019-02-05; First posted 2019-02-22 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Infertility
Keywords: Embryo Transfer; ICSI; Transvaginal Ultrasound
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transvaginal Ultrasound Guided ET (Experimental): Transvaginal ultrasound is used to guide ET
  Interventions: Procedure: Transvaginal Ultrasound Guided ET
- Transabdominal Ultrasound Guided ET (Experimental): Transabdominal ultrasound is used to guide ET
  Interventions: Procedure: Transabdominal Ultrasound Guided ET

INTERVENTIONS:
Procedure: Transvaginal Ultrasound Guided ET — Use of TVUS to guide ET
  Other Names: Transvaginal US guided ET
  Arms: Transvaginal Ultrasound Guided ET
Procedure: Transabdominal Ultrasound Guided ET — Use of TAUS to guide ET
  Other Names: Transabdominal US guided ET
  Arms: Transabdominal Ultrasound Guided ET

SUMMARY:
Randomized controlled study comparing the TVUS versus TAUS guidance during the procedure of embryo transfer.

DETAILED DESCRIPTION:
The aim of this study was to Compare between transvaginal and transabdominal ultrasound guided embryo transfer as regarding clinical pregnancy rate, patient comfort, time required for embryo transfer and endometrial visualization at time of embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing autologous ICSI and frozen embryo transfer (FET) cycles.

Exclusion Criteria:

1. Cases of sever ovarian hyperstimulation requiring embryo cryopreservation
2. Gestational surrogate cycles
3. Oocyte donation cycles
4. Very poor responders
5. Patients with inadequate visualization of the uterus by ultrasound.
6. Very difficult mock embryo transfer.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — A procedure performed only in females
Enrollment: 178 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-03-09 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 3 weeks after Embryo transfer
  A clinical pregnancy is a pregnancy that is confirmed by ultrasonic visualization of gestational sac or heartbeat.

SECONDARY OUTCOMES:
Time required for ET | Time from when the catheter is handed to the transferring physician to the time it is returned to the transferring embryologist.
  Time in seconds required for ET
Degree of cramping and pain | During and immediately after ET
  Degree of cramping and pain from 0 to 10 by visual analogue scale (VAS) where 0 is no pain and 10 unbearable pain.
Endometrial visualization at time of embryo transfer | During ET
  Endometrial visualization at time of embryo transfer by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad S kandil, MD, Study Chair — Menoufia University; Sherif S Gaafar, MD, Study Director — Alexandria University; Haitham A Hamza, MD, Principal Investigator — Menoufia University
Locations (2):
- Egypt (2):
  - Menoufia University, Shibīn al Kawm, Monofiya
  - Alexandria University, Alexandria

IPD SHARING:
Plan to Share IPD: No